CLINICAL TRIAL: NCT03857568
Title: A Phase I, Randomized, Double-blind, Placebo-controlled Study of Intravenous SHR0410 to Evaluate Safety and Pharmacokinetics in Hemodialysis Participants.
Brief Title: A Trial of SHR0410 Injection in Hemodialysis Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR0410-102-AU
Record Dates: First submitted 2019-02-25; First posted 2019-02-28 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR0410 group (Experimental): SHR0410 will be dosed
  Interventions: Drug: SHR0410
- Placebo (Experimental): Placebo will be dosed
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR0410 — drug will be dosed repeatedly
  Arms: SHR0410 group
Drug: Placebo — Placebo will be dosed repeatedly
  Arms: Placebo

SUMMARY:
This is a multi-site study to evaluate the safety and pharmacokinetics of repeated doses of IV SHR0410 in participants who are undergoing hemodialysis.

DETAILED DESCRIPTION:
This is a multi-site study to evaluate the safety and pharmacokinetics of repeated doses of IV SHR0410 in participants who are undergoing hemodialysis. Twenty-four eligible participants will be enrolled into 3 dose cohorts. SHR0410 will be administered after dialysis session. Safety assessments, PK assessments and efficacy evaluations will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study procedures, the risks involved and obtain written informed consent before any study related activity.
* Male or female between the ages of 18 and 75 years, inclusive.
* Male subjects with a partner of childbearing potential must be willing to use a condom when sexually active, throughout the study period and for 28 days following last study drug dosing. Female subjects must be post-menopausal for at least 1 year, permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy) or, if of childbearing potential, must be willing to use a highly effective method of contraception throughout the study period and for 28 days following last study drug dosing.
* Negative drug screen (including alcohol, amphetamines, cocaine, marijuana, opiates, phencyclidine, barbiturates, benzodiazepines, methadone, methamphetamines, tramadol, and tricyclic antidepressants) at screening and on admission to study site.

Exclusion Criteria:

* Anticipated to receive a kidney transplant during the study.
* Known history of allergic reaction to opiates such as hives (Note: side effects related to the use of opioids such as constipation or nausea would not exclude the participants from the study).
* Within 12 months prior to screening, known or suspected history of drug abuse or dependence according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse events in terms of changes in Hematology | 14 days
  Hemoglobin Hematocrit Erythrocytes count Mean cell volume, Mean cell hemoglobin concentration, Leukocytes count, Neutrophils count, Lymphocytes count, Monocytes count, Eosinophils count, Basophils count, Platelets count
Incidence of Adverse events in terms of changes in Urinalysis | 14 days
  Urobilinogen Dipstick urinalysis, including: pH, Specific gravity, Protein, Blood, Leukocytes, Glucose, Ketones, Bilirubin, Nitrites
Incidence of Adverse events in terms of changes in Biochemistry | 14 days
  Including Serum creatinine, Urea, Alanine aminotransferase, Aspartate aminotransferase, Gamma glutamyl transferase, Total bilirubin, Total protein, Albumin, Alkaline phosphatase, Serum uric acid, Glucose, Triglycerides, Total cholesterol, High-density lipoprotein cholesterol, Low-density lipoprotein cholesterol
Incidence of Adverse events in terms of changes in 12-lead ECGs | 14 days
  The 12-lead ECGs must be recorded after the subjects have rested in the supine position for 5 minutes to ensure a stable baseline

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Up to 24 hours post dose
  Plasma SHR0410 Area Under the Concentration-time Curve (AUC)
Time to the peak plasma concentration (Tmax) | Up to 24 hours post dose
  Time to Maximum Plasma SHR0410 Concentration
Peak Plasma Concentration (Cmax) | Up to 24 hours post dose
  Peak Plasma SHR0410 Concentration
Half-time (T1/2) | Up to 24 hours post dose
  Half-time of SHR0410

CONTACTS AND LOCATIONS:
Overall Officials: Neil Boudville, Ph.D, Principal Investigator — Linear Clinical Research Limited
Locations (1):
- Linear Clinical Research, Nedlands, Western Australia(WA), Australia

IPD SHARING:
Plan to Share IPD: No